CLINICAL TRIAL: NCT06557109
Title: PhD, RN Associate Professor
Brief Title: Evaluating the Effects of Popular Music on Cardiopulmonary Resuscitation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gülten Sucu Dağ, PhD, RN Associate Professor, Eastern Mediterranean University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: GSD-1
Record Dates: First submitted 2024-08-02; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: CPR; Training; Music; Nursing Students
Keywords: Cardio-Pulmonary Resuscitation; training methods; music; nursing students

STUDY DESIGN:
Intervention Model Description: randomized posttest control group design
Who Masked: Outcomes Assessor
Masking Description: The evaluator does not know which group is the experimental and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention All students who agreed to participate in the study received theoretical training on Basic Life Support based on the AHA 2015 guidelines from an Emergency Medicine faculty member who holds an AHA First Aid Instructor Certificate for 2 class hours. After the training, the control group students practiced standard CPR, while the intervention group listened to music that would be used during CPR and then performed CPR with music accompaniment.
  Interventions: Other: Popular Music
- Control (No Intervention): Control All students who agreed to participate in the study received theoretical training on Basic Life Support based on the AHA 2015 guidelines from an Emergency Medicine faculty member who holds an AHA First Aid Instructor Certificate for 2 class hours. After the theoretical training, the students were divided into intervention and control groups. After the training, the control group students practiced standard CPR, while the intervention group listened to music that would be used during CPR and then performed CPR with music accompaniment.

INTERVENTIONS:
Other: Popular Music — A funky D mix version of a popular Turkish song
  Arms: Intervention

SUMMARY:
This study aims to analyze short- and long-term effects of musical memory created by using a national popular song on achieving the recommended compression rate and depth and compression-breath rate for nursing students, who received CPR training.

In this study, used a popular Turkish song, entitled, 'More Beautiful Than You' and performed by Duman, to create a musical memory to be used as a mental metronome and analyzed short- and long-term effects of using popular national songs on achieving recommended compression rate and depth and compression-breath rate for nursing students, who received CPR training and performed CPR on high-fidelity simulation mannequins for the first time.

Students in the intervention group practiced CPR with music. Students in the control group practiced CPR with a standard mannequin.

CPR performance of the participants was evaluated just after the CPR training (short-term) and six weeks after the training (long-term).

DETAILED DESCRIPTION:
Nursing students that agreed to participate received two hours of theoretical lecture on basic life support for healthcare professionals.The training was based on the 2015 American Heart Association (AHA) guidelines for CPR and Emergency Cardiovascular Care (ECC) and was provided by an emergency medical expert that had an AHA First Aid Trainer certificate.

Following the theoretical lecture, participants were allocated to the intervention and the control groups and performed at least 5 cycles of CPR (1 cycle=2 minute) on a high-fidelity simulation mannequin at the practice laboratory. During the performance, one of the students delivered rescue breath with a bag valve mask (BVM) whereas the other student performed compression. Participants switched positions after each cycle with 120 compressions.Following the training, students in the control group received the standard CPR training whereas the participants in the intervention group listened to the song to be used in CPR and then performed CPR while listening to the song. CPR performance of the participants was evaluated just after the CPR training (short-term) and six weeks after the training (long-term).

ELIGIBILITY:
Inclusion Criteria:

* third-year nursing students
* who were enrolled in the nursing department
* who did not receive prior CPR training

Exclusion Criteria:

* students that did not agree to participate

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
the primary outcome | CPR performance of the participants was evaluated just after the CPR training (short-term) and six weeks after the training (long-term).
  compression rate of 100-120/min and a depth of 5-6 cm

SECONDARY OUTCOMES:
Secondary outcomes | CPR performance of the participants was evaluated just after the CPR training (short-term) and six weeks after the training (long-term).
  1. arm pain intensity during the CPR Arm pain intensity during the CPR was measured with a 10-cm visual analog scale (VAS).
     Right and Left arm circumference was measured in meters weight in kilograms and height in meters were measured
  2. satisfaction with the CPR training Satisfaction with the CPR training was measured with a 10-cm visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: GULTEN SUCU DAĞ, Last Name, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, North Cyprus Via Mersin, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: Tastan S, Ayhan H, Unver V, Cinar FI, Kose G, Basak T, et al. The effects of music on the cardiac resuscitation education of nursing students. Int Emerg Nurs 2017;31:30-5.
URL: https://pubmed.ncbi.nlm.nih.gov/27406397/

REFERENCES:
- [Result] Tastan S, Ayhan H, Unver V, Cinar FI, Kose G, Basak T, Cinar O, Iyigun E. The effects of music on the cardiac resuscitation education of nursing students. Int Emerg Nurs. 2017 Mar;31:30-35. doi: 10.1016/j.ienj.2016.06.007. Epub 2016 Jul 9. PMID 27406397
- See also: The effects of music on the cardiac resuscitation education of nursing students — https://doi.org/10.1016/j.ienj.2016.06.007